CLINICAL TRIAL: NCT05101343
Title: Use of Fitbits During Breathing Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB21074; P20GM103499-20 (NIH); P217A180094 (Other Grant/Funding Number: Winthrop McNair Scholars Program)
Record Dates: First submitted 2021-09-15; First posted 2021-11-01 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Uses Fitbit, does not participate in breathing meditation.
- Meditation (Experimental): Uses Fitbit and participates in brief, daily breathing meditation.
  Interventions: Behavioral: Breathing meditation

INTERVENTIONS:
Behavioral: Breathing meditation — Daily, 5-minute breathing meditation for one week.
  Arms: Meditation

SUMMARY:
This study will examine short breathing meditations paired with Fitbit technology in order to assess mindfulness and track physical activity. Measures including heart rate, physical activity, sleep patterns, as well as assessments of well-being and anxiety levels, will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Currently a student, faculty, or staff member at university where research is being completed.
* Able to wear a Fitbit close to 24 hours a day for two weeks.

Exclusion Criteria:

* Younger than 18 years.
* Has previously practiced meditation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Guenther, Principal Investigator — Winthrop University - Rock Hill, SC
Locations (1):
- Winthrop University, Rock Hill, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Meditation
Started | 19 | 18
Completed | 17 | 17
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Meditation | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (14) | 31 (13) | 34 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 8 | 18
  Black or African American | 1 | 6 | 7
  Hispanic/Latino/Spanish | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Multi-racial | 2 | 2 | 4
  Prefer not to answer | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Mindfulness
Description: Mindful Attention Awareness Scale (MAAS.) The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness,namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. The survey consists of 15 questions using a Likert scale. Responses range from 1 (Almost Always) to 6 (Almost Never.)The scale is scored by computing a mean of the 15 items on the questionnaire. Score ranges of 15 (low) to 90 (high.) A higher score indicates a higher level of dispositional mindfulness.
Time Frame: Baseline and 2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 17
score on a scale | -0.08 (0.57) | 0.1 (0.43)

2. Primary Outcome: Change in Anxiety
Description: Hospital Anxiety and Depression Scale (HADS). This questionnaire is used to measure anxiety and depression. Scale ranges are from 0 to 3. Lower values represent a better outcome. Total scores for depression and anxiety are summed. A score of 0-7 = normal. A score of 8-10 = borderline abnormal (borderline case.) A score of 11-21 = abnormal (case.)
Time Frame: Baseline and 2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 17
score on a scale | -.18 (2.27) | -2.35 (3.64)

3. Primary Outcome: Change in Well-being
Description: Mental Health Continuum Short Form (MHC-SF.) This questionnaire measures emotional, psychological, and social well-being. It consists of 14 questions scored on a Likert scale ranging from 0-5. Items 1-3 indicate emotional well-being (range 0-15). Items 4-8 indicate social well-being (0-25). Items 9-14 indicate psychological well-being (0-30). Total well-being score as reported here was calculated by adding the three sub-scores together (range 0-70). Higher scores indicate higher well-being for subscales and total well-being.
Time Frame: Baseline and 2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 16
score on a scale | 3.00 (8.89) | 3.75 (10.33)

4. Primary Outcome: Change in Worry
Description: UMC (University Medical Centre) Penn State Worry Questionnaire. This is a 16 item questionnaire. Scale ranges from 0 (Not Typical at All) to 4 (Very Typical.) A higher score indicates a higher propensity for worry.
Time Frame: Baseline and 2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Meditation
Number analyzed (Participants) | 15 | 17
score on a scale | -0.13 (7.03) | -1.59 (6.05)

5. Primary Outcome: Change in Depression
Description: as for outcome 2
Time Frame: Baseline and 2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 17
units on a scale | -1.12 (2.57) | -0.53 (2.90)

6. Secondary Outcome: Change in Sleep Minutes
Description: Duration of sleep in minutes as measured using Fitbit. An increase in duration of sleep indicated improvement.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Duration of sleep in minutes
Arm/Group | Control | Meditation
Number analyzed (Participants) | 14 | 13
Duration of sleep in minutes | -10.76 (36.47) | 6.33 (21.43)

7. Secondary Outcome: Change in Heart Rate
Description: Changes in heart rate in beats per minute as measured by Fitbit (average observed heart rate during Week 2 minus the average heart rate observed during Week 1)
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Beats per minute of heart
Arm/Group | Control | Meditation
Number analyzed (Participants) | 16 | 14
Beats per minute of heart | -0.49 (1.75) | -0.12 (2.84)

8. Secondary Outcome: Change in Steps
Description: Change in number of steps taken as measured by Fitbit (average number of steps taken during Week 2 minus the average number of steps taken during Week 1)
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: number of steps taken
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 15
number of steps taken | -56.12 (1186.91) | 271.96 (1678.45)

9. Secondary Outcome: Change in Physically Active Minutes
Description: Amount of time spent being physically active in minutes as reported by Fitbit. An increase in time spent being physically active indicated improvement.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Duration of physical activity minutes
Arm/Group | Control | Meditation
Number analyzed (Participants) | 17 | 15
Duration of physical activity minutes | -7.45 (33.45) | 3.02 (49.7)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 weeks
Description: 34
Arm/Group | Control | Meditation
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT05101343/Prot_SAP_000.pdf